CLINICAL TRIAL: NCT05094115
Title: Enhancing Resiliency and Optimizing Readiness in Military Personnel
Acronym: R2OE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC20210486H; W81XWH-19-1-0628 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Resilience, Psychological; Stress, Physiological
Keywords: Psychological flexibility

STUDY DESIGN:
Intervention Model Description: All participants will receive usual training with randomized participants being assigned to psychological flexibility training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training as usual (No Intervention): Training as Usual for the 3rd SFAB is the U.S. Army Master Resilience Trainer (MRT). It focuses on teaching resilience skills and is one of the foundational pillars of the Comprehensive Soldier Fitness program. MRT course is intended to impart training resilience skills, designed to introduce other resilience concepts that soldiers will likely encounter through their careers. Key focus of course are (1) resilience, (2) building mental toughness, (3) identifying character strengths, and (5) strengthening relationships. The 3rd SFAB uses a a team training grounded in strengths-based leadership. The Small Team Development Consultant and Brigade Behavioral Health Provider serves as a consultant to units conducting their own resiliency training as usual. No booster sessions will be offered to Training as Usual.
- Training as usual with psychological flexibility training (Active Comparator): Training as usual, with psychological flexibility training delivered during a 2-day workshop.
  Day 1 provides an overview of the training and describes the posture or stance to prepare for response to challenging situations in a psychologically flexible manner.
  Day 2 provides common coping strategies.
  Interventions: Behavioral: Psychological Flexibility Training (PFT)

INTERVENTIONS:
Behavioral: Psychological Flexibility Training (PFT) — A 2-day workshop lasting approximately 8 hours per day. Day 1: an overview of the training and to describe the posture or stance that prepares one to respond to challenging situations in a psychologically flexible manner.
  Day 2: identifies common coping strategies that typically fail or even "backfire" over the long term and to practice skills that promote psychological flexibility. Experiential exercises will be integrated throughout the training.
  Following the PFT, 4 optional, monthly, one-hour booster sessions to supply refresher information.
  * An experiential exercise to highlight one or more process/concept that was introduced during the 2-day training.
  * Questions from the attendees about applying the concepts in their lives.
  * Comments and questions from the booster session facilitators to encourage application of the concepts.
  Arms: Training as usual with psychological flexibility training

SUMMARY:
Security Force Assistance Brigades (SFABs) are specialized United States Army units formed to train, advise, assist, enable and accompany operations with allied and partner nations. Security Force Assistance Brigades are composed of roughly 800 senior military personnel, primarily commissioned and non-commissioned officers selected from regular Army units across a wide range of military specialties. Because of the high operational tempo (OPTEMPO) of these units, individual resiliency is of utmost importance in maintaining readiness to successfully execute critical, high-stress missions. Acceptance and Commitment Training (ACT) is an evidence-based intervention with strong potential to enhance resiliency by bolstering psychological flexibility along with other factors which have been demonstrated to optimize individual and group performance. This project will compare an Acceptance and Commitment Training-based resiliency-enhancement training program as compared to training as usual in 600 3rd Security Force Assistance Brigades soldiers stationed at Fort Hood in Killeen, Texas. Assessment measures related to resilience will be administered before and after training as well as before and after deployment. Assessments will be conducted at baseline, and every 4 months thereafter for a total of 16-months.

DETAILED DESCRIPTION:
Over the past decade, the Department of Defense has also had a significant interest in the development and evaluation of evidence-based programs for enhancing resiliency in military personnel to help optimize operational readiness and prevent deployment-related psychological health causalities (Peterson, Cigrang, & Isler, 2009). Maintaining health, optimizing performance, and boosting resiliency to stressors in harsh combat environments is a momentous challenge. Conducting research aimed at enhancing health, performance, and resiliency is similarly challenging. As a result, few studies have documented evidence-based interventions to maintain or boost performance under such harsh conditions. Thus, compared to the major scientific and clinical advancements in the assessment and treatment of deployment-related psychological health conditions in active duty military personnel, little research has been conducted on the enhancement of resiliency in military personnel. A major challenge in the development and evaluation of evidence-based resiliency-enhancement programs for military personnel is the design of scientifically valid and methodologically sound research designs. Most of the resiliency-enhancement programs developed to date-such as the Comprehensive Soldier Fitness Program-have been evidenced-informed programs that were universally implemented in ways that prevented rigorous scientific validation of their efficacy (Steenkamp, Nash, & Litz, 2013). Consequently, prospective efficacy research is desperately needed to evaluate potential approaches to enhance resiliency and optimize readiness in military personnel.

Ideally, a resiliency enhancement training for military personnel would demonstrate not only improvements in self-reported resiliency and other related constructs but also demonstrate positive adaptation in the face of significant stress or adversity as a result of the training (Britt, Sinclair, & McFadden, 2013). Adler and colleagues have conducted a series of studies to evaluate the efficacy of resiliency training in active duty military populations (Adler, et al., 2015; Adler et al., 2015; Cacioppo et al., 2015).

An excellent summary of the science of resiliency was completed as part of a systematic review by Macedo et al., (2014) of interventions for building resilience in non-clinical samples of adults. The summary of this review highlighted that to date, no prospective study has evaluated the efficacy of resiliency-enhancement trainings and investigated the actual occurrence of adverse situations after the training to document that the training improved positive adaptation in the face of significant adversity. A Cochrane Report titled Psychological Interventions for Resilience Enhancement in Adults (Helmreich et al., 2017) is currently conducting a comprehensive review of the scientific literature on psychological interventions to enhance resiliency in adults. The currently published protocol for this Cochrane study indicates that Acceptance and Commitment Therapy is one of the most promising psychological approaches for resilience enhancement in adults. The study team believe that Acceptance and Commitment Therapy has some of the strongest scientific support for potential adaptation for use in military training to enhance resiliency and optimize readiness.

Acceptance and Commitment Therapy, which is pronounced as one word ("act"), is a contemporary, evidence-based, cognitive-behavioral approach to improving functioning and performance (Hayes, 2004; Hayes et al., 2006). In Acceptance and Commitment Therapy, the broad goal is to help individuals identify and act consistently with their values and goals and to align their actions with those values even if they are experiencing pain or discomfort (Hayes, 2004; Hayes et al., 2006). Acceptance and Commitment Therapy is rooted in a well-established theory of human language and cognition (Relational Frame Theory), which describes how internal experiences (e.g., thoughts, emotions, physiological sensations, and urges) are viewed as behaviors that can be predicted and influenced. In Acceptance and Commitment Therapy, trainees practice identifying these internal events for what they are (i.e., transient phenomena) rather than as permanent experiences. Trainees learn to take a stance characterized by active acceptance of and willingness to remain in contact with these experiences rather than allocating attention and energy to attempts to control, reduce, or eliminate negatively evaluated internal experiences. Examples of such negatively evaluated internal experiences include physiological sensations such as pain or sensations associated with lack of oxygen, emotions such as fear, and thoughts such as "I can't stand it" or "It's not worth it." Under harsh conditions, it is highly unlikely if not impossible that attempts to control, suppress, or eliminate such experiences will be successful. Thus, a behavioral stance characterized by active acceptance and willingness is more adaptive, as it increases the availability of personal resources for optimizing volitional control over one's behavior. This volitional control may then be optimally applied toward goal attainment. Taking an accepting, willing stance ultimately gives rise to greater psychological flexibility, which is the primary target or mechanism in Acceptance and Commitment Therapy. As with elite athletics, taking an adaptive, flexible stance is a core element of preparation for successful performance.

There are over 250 published or in press randomized controlled trials (RCTs) using Acceptance and Commitment Therapy to optimize functional outcomes in diverse domains including improving workplace performance under stressful conditions, completing physical exercise regimens, improving parenting skills, and adhering to dietary restrictions (Moran, 2015). Moreover, Acceptance and Commitment Therapy has been studied extensively and demonstrated to improve functioning among people living with a wide range of psychological and physical conditions, syndromes, and injuries. Such randomized controlled trials span applications of Acceptance and Commitment Therapy for depression, anxiety disorders, substance use disorder, psychosis, personality disorders, tobacco use, eating disorders, and a range of medical health issues (e.g., cancer, diabetes, chronic pain). Thus, Acceptance and Commitment Therapy has a proven track record of improving performance and functioning across a range of conditions, including those involving intense physical and emotional distress.

According to the Acceptance and Commitment Therapy model, suffering and impairment are primarily the consequence of psychological inflexibility (i.e., inability to persist in or change behavior according to situational or contextual factors and personally chosen values due to problematic, inflexible reactions to negatively evaluated internal experiences). Psychological inflexibility may be particularly detrimental when an individual is confronted with stress or adversity (Hayes, 2004; Hayes et al., 2006). Thus, interventions targeting increased psychological flexibility-Acceptance and Commitment Therapy being the foremost in this field-are recommended not only for facilitating recovery after stressors but also for enhancing resilience (e.g., Meyer, Frankfurt, et al., 2018; Meyer, Szabo, et al., 2019). Highly relevant to the current proposal is a series of randomized experiments in which brief interventions based on core components of the Acceptance and Commitment Therapy model were shown to increase pain tolerance. In these studies, pain tolerance was operationalized as increasing the amount of time spent on the task before quitting, which is an analogue for greater persistence in an intense military training program. A brief acceptance-based intervention led to large increases in pain tolerance compared to a control group (Masedo & Rosa Esteve, 2007). Recently, a brief values-based intervention led to a 55% increase in pain tolerance, whereas the control condition reported a 12% decrease in pain tolerance at follow-up (Smith et al., 2018).

Additional empirical support for the Acceptance and Commitment Therapy model comes from a study led by Co-PI Meyer demonstrating that psychological flexibility predicted lower overall disability and greater quality of life in combat-exposed veterans, even after accounting for Post Traumatic Stress Disorder symptom severity (Meyer, Frankfurt, et al., 2018). Acceptance and Commitment Therapy includes mindfulness training to support the development of psychological flexibility. This same study also found that mindfulness predicted lower disability and greater quality of life in combat veterans over and above Post Traumatic Stress Disorder severity. In Acceptance and Commitment Therapy, these modifiable factors are targeted in order to promote trainees' ability to commit to engaging in goal- or values-consistent behavior.

Consistent with the Acceptance and Commitment Therapy model, the recent report by the Cochrane Collaboration that identified Acceptance and Commitment Therapy as an evidence-based intervention for enhancing resilience listed psychological flexibility, the central target of Acceptance and Commitment Therapy, as having the highest tier of evidence support for promoting resilience (Helmreich et al., 2017). They also rated this relationship as having the highest tier of empirical support. Specifically, more systematic reviews and meta-analyses were included in the report for psychological flexibility than any other single factor. The report delineated how Acceptance and Commitment Therapy is likely to enhance resilience by bolstering psychological flexibility specifically through teaching mindfulness and acceptance skills (e.g., maintaining contact with the present moment, cognitive de-fusion, acceptance of or willingness to experience emotional distress) along with behavior-change skills (e.g., committed action). In this way, the report authors posit several resilience factors will be fostered in Acceptance and Commitment Therapy-based resilience interventions (e.g., cognitive flexibility, purpose in life). In particular, based on the available evidence, the report emphasized that acceptance of the full range of emotions, particularly those that are uncomfortable and that is often associated with behavioral avoidance, likely promotes successful adaptation to stressful conditions (i.e., resilience; Helmreich et al., 2017).

Security Force Assistance Brigades are specialized United States Army units formed to train, advise, assist, enable and accompany operations with allied and partner nations. SFABs are intended to reduce the burden of such operations on conventionally organized Brigade Combat Teams (BCTs), allowing Brigade Combat Teams to focus on fighting near-peer threats. Designed on the model of a standard infantry Brigade Combat Teams, Security Force Assistance Brigades is composed of roughly 800 senior personnel, primarily commissioned and non-commissioned officers selected from regular Army units and given additional training at the Military Advisor Training Academy at Fort Benning, Georgia. The first such unit, the 1st Security Force Assistance Brigades, began operations in February 2018. The 3rd Security Force Assistance Brigades began operations at Fort Hood less than a year later in January 2019.

As with other highly trained and specialized military units deployed to hostile and uncertain areas, the 3rd Security Force Assistance Brigades has been and will continue to be exposed to physical and psychological stressors as part of their military service.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 or older
* Male or female soldiers assigned to the 3rd SFAB

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale (CD-RISC) | Baseline to 16 months
  Change in score on a 10-item questionnaire examining attitudes toward coping with adversity. Items require respondents to indicate their degree of endorsement on 5-point scales ranging from 0 ("not true at all") through 4 ("true nearly all the time"; e.g., "Having to cope with stress makes me stronger"). Score ranges are from 0 to 40, with a lower score indicating less coping ability.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Peterson, PhD, Principal Investigator — University of Texas Health San Antonio
Locations (1):
- Fort Hood, Killeen, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in the STRONG STAR Repository and available to other researchers upon request and approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the completion of the study and publication of main outcomes for a minimum of 5 years.
Access Criteria: Requests for access to the data can be emailed to repository@strongstar.org.

REFERENCES:
- [Derived] Peterson AL, Moore BA, Evans WR, Young-McCaughan S, Blankenship AE, Straud CL, McLean CS, Miller TL, Meyer EC; STRONG STAR Consortium. Enhancing resiliency and optimizing readiness in military personnel through psychological flexibility training: design and methodology of a randomized controlled trial. Front Psychiatry. 2024 Jan 5;14:1299532. doi: 10.3389/fpsyt.2023.1299532. eCollection 2023. PMID 38250282